CLINICAL TRIAL: NCT02249286
Title: Child-Centred Counselling and Home-Based Food Production to Improve Dietary Adequacy and Growth of Young Children in Southwest Ethiopia
Brief Title: Integrating Nutrition Education & Household Food Production for Child Nutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jimma University (Other)
Collaborators: Nestlé Foundation (Other); Flemish Interuniversity Council (VLIR) (Network)
Responsible Party: Principal Investigator, Abebe Gebremariam, Professor, Jimma University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCC-HFP
Record Dates: First submitted 2014-09-05; First posted 2014-09-25 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: Behavior
Keywords: Child Centered Counseling; Home based food production; Nutrition; Health; IYCF
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Child Centered Nutrition Counseling (Experimental): The intervention comprises child-centered nutrition counseling for caretakers and support for 'developed' gardens and improved backyard poultry production.
  Interventions: Behavioral: Child Centered Nutrition Counseling; Other: no intervention
- No intervention (No Intervention)

INTERVENTIONS:
Behavioral: Child Centered Nutrition Counseling — The intervention comprises child-centered nutrition counseling for caretakers and support for 'developed' gardens and improved backyard poultry production; whereas the control will only receive the agriculture extension and the existing health and nutrition education in the area
  Arms: Child Centered Nutrition Counseling
Other: no intervention — the control will only receive the agriculture extension and the existing health and nutrition education in the area
  Arms: Child Centered Nutrition Counseling

SUMMARY:
In Ethiopia, a child-centered counseling approach is hypothesized to be more effective than the current nutrition and health education when investment on home-based food production is used as a platform for nutrition education. This project is proposed to evaluate the efficacy of a food-based package integrating child-centered nutrition counseling and home-based food production using a between-group comparative intervention study. The intervention comprises child-centered nutrition counseling for caretakers and support for 'developed' gardens and improved backyard poultry production.

DETAILED DESCRIPTION:
Growth faltering among Ethiopian infants and young children is one of the highest in sub-Saharan Africa. Nutrition education on infant and young child feeding has shown good potential to improve growth of young children whenever it is accessible, context-based and integrated with locally available resources. The current nutrition education in Ethiopia, however, appears to be general and lacks the essential components for success. It is mainly didactic and lacks a motivational approach that can enhance the self-efficacy of mothers for behavior change. Another important barrier for nutrition education to become effective is that rural mothers have limited access to nutrient-dense foods that are recommended to be fed to young children. Therefore, it is expected that low food access by poor households together with the less motivational approach used may hamper the effectiveness of the current nutrition education in the country. In Ethiopia, a child-centered counseling approach is hypothesized to be more effective than the current nutrition and health education when investment on home-based food production is used as a platform for nutrition education. This project is proposed to evaluate the efficacy of a food-based package integrating child-centered nutrition counseling and home-based food production using a between-group comparative intervention study. The intervention comprises child-centered nutrition counseling for caretakers and support for 'developed' gardens and improved backyard poultry production; whereas the control will only receive the agriculture extension and the existing health and nutrition education in the area. Two Primary Healthcare Units (one intervention and one control group) will be selected from Jimma Zone using relevant criteria. A total of 404 (i.e. 202 in each of intervention and control areas) households with infants of age < 12 months will participate in the study for 18 months. The efficacy of the intervention will be assessed by its effect on child growth and infant and child feeding index as primary outcomes. Besides the effect on dietary adequacy and growth, the project aims at evaluating the interactive processes in a longitudinal way to provide evidence on the possible success factors and barriers encountered. Therefore, secondary outcomes include household production, income and expenditure in relation to the home-based food production; diet diversity; feeding and care practices, and morbidity. Data will be compared between intervention and control groups using linear mixed-effects models and generalized linear models.

ELIGIBILITY:
Inclusion Criteria:

* infants less than 12 month
* are permanent residents in the area;
* have no plan to move away during the intervention period;
* are willing to adopt the agriculture activities; and
* have adequate place and time to adopt developed gardens & backyard poultry production

Exclusion Criteria:

* infants with severe acute malnutrition warranting referral to nutrition rehabilitation program with Ready-To-Use Therapeutic foods
* severely ill infants with clinical complications warranting hospital referral; and
* infants with obvious congenital or chronic abnormalities that impair feeding or physical growth measurements.

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 404 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Child growth [-Prevalence of stunting ][<-2SD] | baseline,18 month
  prevalence of stunting will be determined by height for age (Ht/Age) using height /length measured in the recumbent position to the nearest 0.1 cm using a measuring board with an upright wooden base and movable headpiece. as well actual age of child will be taken and expressed in terms of Z score.

CONTACTS AND LOCATIONS:
Overall Officials: Abebe Gebremariam, Professor, Principal Investigator — Jimma University; Alemayehu Argaw, Mr, Principal Investigator — Jimma University; Lieven Huybregts, Dr, Principal Investigator — University Ghent; Patrick Kolsteren, Professor, Principal Investigator — University Ghent; Mulusew Gerbaba, Mr., Principal Investigator — Jimma University; Solomon Demeke, Professor, Principal Investigator — Jimma University; Joep Grosemans, Mr., Principal Investigator — Provincial university college Limburg; Amanuel Tesfay, Mr., Principal Investigator — Jimma University